CLINICAL TRIAL: NCT02069431
Title: Effects of Oxytocin on Physical and Cognitive Functioning in the Elders
Brief Title: Oxytocin Aging Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was halted prematurely due to the COVID-19 pandemic, resulting in the inability to enroll participants. Funding for this project has also ended.
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201300801-N; AG028740 (Other Grant/Funding Number: Pepper Center); P30AG028740 (NIH); F016327 (Other Grant/Funding Number: UF FOU); AGR DTD 09-01-2016 (Other Grant/Funding Number: Price-IOA-CTSI)
Record Dates: First submitted 2014-02-10; First posted 2014-02-24 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Inflammation
Keywords: inflammation; physical function; cognitive function
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Oxytocin spray (Experimental): Intranasal OT (24 IUs) self-administration will take place twice a day over a 28-day period.
  Interventions: Drug: Intranasal Oxytocin spray
- Intranasal Placebo spray (Placebo Comparator): placebo (containing all of the inert ingredients except for the oxytocin) self-administration will take place twice a day over a 28-day period.
  Interventions: Other: Intranasal Placebo spray

INTERVENTIONS:
Drug: Intranasal Oxytocin spray — Intranasal OT (24 IUs) self-administration will take place twice a day over a 28-day period.
  Arms: Intranasal Oxytocin spray
Other: Intranasal Placebo spray — placebo (containing all of the inert ingredients except for the oxytocin) self-administration will take place twice a day over a 28-day period.
  Arms: Intranasal Placebo spray

SUMMARY:
The life expectancy of older Americans continues to increase, with persons aged > 65 years representing the fastest growing segment of the US population (Manton et al., 1995). While prolongation of life remains an important public health goal, a goal of even greater significance is that extended life should involve preservation of the capacity to live independently and to function well physically, cognitively, and socioemotionally (Katz et al., 1983). Therefore, identification of proven interventions to maintaining functioning across these domains and prevent disability is a major public health challenge (Branch et al., 1991). Greater physical and cognitive independence in older adults has been shown to crucially influence social integration in old age (Cornwell & Waite, 2009), resulting in significant increase in quality of life and reduction of risk for morbidity and mortality, social stress, anxiety, and depressive symptoms (Bassuk et al., 1999; Seeman, 1996). A promising candidate to promote functional levels across physical, cognitive, and socioemotional domains is the neuropeptide oxytocin (OT) (Barraza et al., 2013; Bartz et al., 2011; Feifel et al., 2012; Meyer-Lindenberg et al., 2011; Szeto et al., 2012). Combining neuroendocrine with behavioral approaches (e.g., performance-based measures of physical and cognitive function), the proposed multidisciplinary research therefore sets out to clarify the extent to which intranasal administration of OT over a period of 4 weeks can reduce inflammation and improve physical and cognitive function in older men. Constituting a complementary piece to the IRB approved currently ongoing Faces Study (IRB # 39-2013), this project will also allow examination of interactions between OT's effect on physical health, cognition, and socioemotional function.

DETAILED DESCRIPTION:
Overview:

* Initial screening visit
* 3 baseline study visits
* 4-week treatment phase
* 3 study visits after treatment
* Follow-up phone contact

All study visits will be conducted at the Institute on Aging or the McKnight Brain Institute at the University of Florida. The treatment phase will take place in the participant's home.

The participant will be assigned by chance to receive either the oxytocin or the placebo. The placebo is a substance, like salt water, that looks like and is given in the same way as the oxytocin but contains no oxytocin. Neither the participant nor the research assistant will know which type of dose they are getting. This information is coded and securely stored away until the data is analyzed, but that information is available if it is needed.

Screening Visit: Together with the information obtained in the phone pre-screening that the investigators have already conducted, the main purpose of the screening visit is to find out if the participant is eligible to participate in the study.

* The investigators will ask the participant questions about their health condition and recent activities and the investigators will review the participant's current and past medical health as well as their education and living situation.
* The participant will then have a short physical exam by a licensed physician including measurement of blood pressure and pulse, and a brief consultation to go over the participant's medical review. This will not be a clinical doctor visit for routine medical care, but a visit to confirm the participant's eligibility to participate in the study. Next, the participant's vision will be tested. The participant will be asked to view a rotating C-shape and identify the direction of the break in the C faces. The C will get larger and smaller depending on the participant's response and in another task the shade of grey for the C and the background will vary.

Then the physical status of the participant will be determined based on the following activities:

* The participant will be asked to walk at his/her usual pace for a distance of 13 feet (4 meters) two (2) separate times.
* The participant will be asked to stand from a sitting position, without using their arms. If they are able to perform this task, they will be asked to stand up from and sit down on a chair five (5) times as fast as they can.
* The participant will be asked to maintain their balance while standing in three different positions, 1) with feet together, 2) with the heel of one foot beside the big toe of the other foot, and 3) the heel of one foot in front of and touching the toes of the other foot.
* A blood draw (~30milileters or ~2 tablespoons) and urine collection (~2mL or ~0.14 tbs) will follow. Result of blood or/and urine testing may indicate that the participant should not participate in the study. The blood test will also be used to determine the level of oxytocin occurring normally in the participant's blood and to determine level of inflammation in their body. If any incidental or clinically significant findings occur, the investigator will inform you of this and give you a copy of the lab results. The participant will also be encouraged to see their primary care physician.
* Some of the blood and a saliva sample (~2mL or ~ 0.14 tbs) that the participant will be asked to provide will help to find out how the activity of their genes may impact how they perform on some tests. All samples will be stored in a locked space at the Institute on Aging.

Baseline Visit 1:

* The investigator will ask the participant to engage in a series of tests and answer questionnaires related to physical, auditory (hearing), and social and emotional functioning.
* The first test is a learning and remembering task.

This is followed by a Physical Test Battery:

* The participant will be asked to walk for 6 minutes.
* The participant will also be asked to walk a distance of 33 feet (10 meters) three times. They will be asked to walk the same distance another three times while counting out loud.
* The participant will be asked to perform upper- and lower-body muscle strength and endurance assessment
* The participant will be asked to respond to various questionnaires related to their physical health.

Auditory Test Battery o The participant will be asked to complete tasks that require them to listen and attend to desired stimuli in the presence of a competing message or noise.

Socioemotional Test Battery

o The participant will be asked to complete questionnaires to measure their social and emotional health, which will include questions to measure their current mood, their general level of trust, their level of loneliness, and their drive to identify emotions and thoughts in others and to respond to these with an appropriate emotion. These questions will also measure the participant's selflessness and concern for the well-being of others, their emotional attention and clarity, their anxiety level, and personality.

Baseline Visit 2:

* At the beginning of this visit, we will ask the participant about recent activities.
* The participant will then be asked to participate in an electroencephalography (EEG) recording session, that is a recording of electrical activity along their scalp. An EEG cap, selected for the participant's head size, will be placed on their head. The cap contains small electrodes that record brain electrical activity. During this part of the study, the participant will sit in a chair while watching pictures on a computer screen and listening to sounds through headphones, or resting.
* While recording EEG, the participant's eye movements will be monitored with an eye tracker. The eye-tracking camera will be placed in front of them and after a brief calibration procedure will track the participant's eye movements while viewing stimuli on the screen and hearing sounds.
* Before the tasks start, the participant will receive detailed information and have a chance to ask any questions that they may have about the tasks or about the EEG and eye tracking procedures. The participant will also have the chance to work on some practice trials.
* After the EEG and eye tracking recording, the investigator will then ask the participant about the amount of pain they experienced in the last 6 months.
* This will be followed by brief sensory testing. In particular, the investigator will apply pressure to several sites on the participant's face and body. The pressure will be slowly increased, and the participant will be asked to tell the investigator when they begin to feel discomfort or mild pain. As soon as the participant indicates that they feel pain, the pressure will be removed. Also, the investigator will tap the participant with a small nylon tip on their knee and the back of their hand and will ask the participant to indicate how painful this feels. The investigator will do that twice at each site.

Baseline Visit 3:

* At the beginning of this visit, the investigator will ask the participant about their recent activities.
* If the participant is assigned to the MRI/MRS portion of the study the investigator will ensure that they are eligible and safe to participate in the scanning session that day.
* The participant will then practice the tasks that they will work on while in the MRI scanner. The tasks will involve viewing geometrical shapes, faces, and images of objects and scenes. The participant will receive detailed information and have a chance to ask any questions that they may have about the tasks or about the MRI procedure before they go into the scanner.
* At this point, the participant will be shuttled to the McKnight Brain Institute, and get settled into the MRI scanner, all with the assistance of the trained researcher.
* While the participant is resting comfortably in the scanner, the investigator will ask them to work on the tasks mentioned above and while they do the MRI machine will produce images of their brain, as well as scan their brain at rest. The participant will be in the scanner for less than 60 minutes.
* The investigator will ask the participant to engage in a series of tests and respond to questionnaires related to their memory and thought process.
* This Cognitive Test Battery comprises:
* Tasks that ask the participant to attend to, respond to, or remember various stimuli on the computer screen and on paper.

Intervention Phase:

* The participant will self-administer either oxytocin or a placebo into their nose by using a nasal spray bottle. The spray will be administered twice a day over 4 weeks. The investigator will give the participant guidance about how to administer the spray and will ask them to keep a log book of their oxytocin/placebo administration.
* In addition, during the treatment phase the investigator will ask the participant to fill in a short diary about social activities they engaged in during their day as well as emotions they experienced.
* In Week 1 and 4 of the intervention phase, the participant will be fitted with a device (i.e., bio-harness) that allows the investigator to measure physiological functions of the participant's body such as their heart rate and breathing rate, for over a period of 24 hours while the participant engages in their daily activities. The participant will be asked to wear it on a typical day, representative of their normal daily activity. The 24-hour period will be one in which the participant is not traveling out of town. A trained research assistant will visit the participant in their home to fit them with and take off the bio-harness. The bio-harness will be comfortably fitted with a chest strap around the participant's upper body. It generally will not affect the clothes the participant can wear, it is water resistant, and the participant will be able to pursue the large majority of their daily activities in the usual manner.
* During the treatment phase, research assistants will call the participant once a week to ask whether they experience any drug side effects or any problem with their health.

Post-Treatment Visit 1:

* The investigator will ask the participant questions about their health condition and recent activities.
* The participant will again be physically examined (including vitals) under the supervision of a licensed physician.
* Another blood draw (~30mL or ~2 tbs) will be conducted to run blood tests and determine the level of oxytocin after the treatment phase as well as the level of inflammation in the participant's body. Urine (~2mL or ~0.14 tbs) will be collected again to ensure that no adverse changes have occurred during the treatment phase. The samples will be stored in a locked space at the Institute on Aging.
* The investigator will again ask the participant to engage in a series of tests and respond to questionnaires related to recent activities as well as physical, auditory (hearing), and their social and emotional functioning. These measures will be very similar to the ones they did before the intervention phase.

Post-Intervention Visit 2:

* At the beginning of this visit, the investigator will ask the participant about recent activities.
* The investigator will ask the participant to participate in ERP and eye tracking recordings similar to the ones before the treatment phase.
* The investigator will also ask the participant to engage in a series of tests and respond to questionnaires related to their memory and thought process. These measures will be very similar to the ones they did before the treatment phase.
* This will be followed by brief sensory testing, similar to the one that took place before the treatment phase.

Post-Intervention Visit 3:

* At the beginning of this visit, the investigator will ask the participant about recent activities.
* If the participant is assigned for the MRI/MRS portion of the study the investigator will ensure that the participant is eligible and safe to participate in the scanning session that day.

The participant will then practice the tasks that they will work on while in the MRI scanner, which will be similar to the ones they engaged in before the treatment phase.

* At this point, the participant will be shuttled to the McKnight Brain Institute, and get settled into the MRI scanner, all with the assistance of the trained researcher.
* The participant will again be in the scanner for less than 60 minutes.
* The investigator will ask the participant to engage in a series of tests and respond to questionnaires related to their memory and thought process, similar to the ones they engaged in before the treatment phase.
* Upon completion of the study, the investigator will tell the participant about the general goals of the study and answer any questions that they may have

  1-Week Follow-Up Phone Call:
* A research assistant will call the participant about one week after the participant's last study visit to inquire whether they experienced any drug side effects or any health problems.

The genetic material that is obtained from the blood, saliva, and urine samples will be stored until the end of the study. By temporarily storing the genetic material, the investigator will be able to examine the importance of different oxytocin genes as well as other genes that are not yet known as being involved in how people think and behave.

When there is no longer sufficient amounts of blood, saliva, and urine samples for analysis, or samples become degraded, or the participant requests in writing that the sample be destroyed, any remaining genetic material will be destroyed. The genetic material will only be accessible to the research staff and will be labeled only by an identification number, not the participant's name. The University of Florida will not sell the samples and will not use the DNA for cloning.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 55 years or older
* generally healthy physically and cognitively
* blood pressure < 180/100 mm Hg
* willing and able to give informed consent.

Exclusion Criteria:

* participants will be extensively screened for study eligibility aligning with study and safety requirements related to drug application and Magnetic Resonance Imaging (MRI)/Magnetic Resonance Spectroscopy (MRS)

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-02; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
The use of intranasal oxytocin (OT) will reduce inflammatory biomarkers in older men and women after the 4 week treatment (post intervention). | Day 28
  The use of intranasal OT will reduce inflammatory biomarkers (IL-6, tumor necrosis factor (TNF)-α, TNF-sR1, TNF-sR2, CRP) measured in blood samples.

SECONDARY OUTCOMES:
The use of intranasal OT will improve objective and subjective physical function (gait, balance, fatigue, etc.) in older men and women after the 4 week treatment (post intervention). | Day 28
The use of intranasal OT will improve socioemotional function (face processing, emotion processing, etc.) in older men and women after the 4 week treatment (post intervention). | Day 28

OTHER OUTCOMES:
The use of intranasal OT will improve auditory and cognitive function (executive functioning, attention, memory, etc.) in older men and women after the 4 week treatment (post intervention). | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Natlie Ebner, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Clinical Research Center, Gainesville, Florida
  - UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida